CLINICAL TRIAL: NCT03882086
Title: Randomized Controlled Trial Of The Effect Of Foot Reflexology On Sleep Quality Of Postpartum Women
Brief Title: Foot Reflexology on Postpartum Sleep Qualıty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ilkay Arslan, Assoc. Prof. Dr., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2019-03-10; First posted 2019-03-20 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Postpartum Women
Keywords: Foot reflexology; nursing; postpartum period; postpartum sleep quality

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot reflexology group (Experimental): The intervention group was comprised of 30 women in the early postpartum period. Pretest data were collected on the 14th day postpartum. Then a total of four reflexology sessions were applied for 15 minutes in each foot, in the afternoons, every other day between postpartum 14th-20th day, as the women were available. And posttest data were collected on the 20th day postpartum at the end of the four-reflexology sessions.
  Interventions: Other: foot reflexology
- standard care group no reflexology (No Intervention): The control group of this study was comprised of 30 women in the early postpartum period who had sleep problem and gave vaginal birth. Pretest data were collected on the 14th day postpartum. On the 20th day postpartum, the posttest data were assessed during home visits. These women only received routine postpartum care from public health nurses but did not access the reflexology

INTERVENTIONS:
Other: foot reflexology — Four sessions foot reflexology was applied for 15 minutes in each foot, every other days between postpartum 14th- 20th day
  Arms: foot reflexology group

SUMMARY:
Aim and objectives: To determine the efficacy of foot reflexology versus standard care for improvement of the sleep quality of postpartum women following vaginal birth.

Background: Sleeplessness is one of the major problems experienced by women in the postpartum period following vaginal birth.

Design: A single-blind, randomized controlled trial was conducted between July 2016 and March 2017.

Methods: In this trial, a total of 54 postpartum women were divided into the intervention group (n= 24) and control group (n= 30). In the intervention group, four sessions foot reflexology was applied for 15 minutes in each foot, every other days between postpartum 14th- 20th day. Measures included daily and nighttime sleep durations and Postpartum Sleep Quality Scale (PSQS) scores. This study was used the CONSORT scheme.

DETAILED DESCRIPTION:
This study was a single-blinded, randomized controlled trial with a prospective pretest-posttest experimental design. This study was conducted between July 2016 and March 2017. Postpartum women were visited at their homes following vaginal birth in the obstetrics clinic of XXX State Hospital in Turkey.

To calculate the sample size, we utilized a 95% confidence interval, 80% power, and a 0.8 effect size. Accordingly, the sample size was determined to be 60 (30 control, 30 intervention) as calculated a priori with a t test using G Power package software. The study was completed with 54 women due to some of the women dropping-out of the study, with 24 women in the intervention group and 30 women in the control group. In this study, the simple randomization method (Statistical Analysis System Institute, Cary, North Carolina, version 8.2) was used to create an equal number of samples in both groups. Thus, participants were single-blinded to treatment allocation. Also the first researcher delivered the intervention and, therefore, could not be blinded to allocation. This study was used the CONSORT scheme.

A total of four reflexology sessions were applied in the afternoons every other day between postpartum days 14 through 20. Pretest data were collected on the 14th day and posttest data were collected on the 20th day. This pilot study revealed that no changes were required in the study method. The five women who participated in the pilot study were excluded from the study data.

The intervention group was comprised of 30 women in the early postpartum period. Pretest data were collected on the 14th day postpartum. Then a total of four reflexology sessions were applied for 15 minutes in each foot, in the afternoons, every other day between postpartum 14th-20th day, as the women were available. And posttest data were collected on the 20th day postpartum at the end of the four-reflexology sessions.

The control group of this study was comprised of 30 women in the early postpartum period who had sleep problem and gave vaginal birth. Pretest data were collected on the 14th day postpartum. On the 20th day postpartum, the posttest data were assessed during home visits. These women only received routine postpartum care from public health nurses but did not access the reflexology.

Data were collected by Personal Information Form and Postpartum Sleep Quality Scale. Data were evaluated using SPSS-17 software (Statistical Package for Social Sciences). Descriptive data were expressed as score means, standard deviations, and min-max values, and normal distribution was measured with kurtosis and skewness. The t test and Mann Whitney U test (z) were used to determine the significance of the differences between pretest and posttest sleep duration and quality in the control and intervention groups according to the hypotheses. Values of p < 0.05 were considered significant. Due to the dropouts in the intervention group, an Intention to Treat (ITT) analysis was performed. Mean method was used with the mean of the sample followed for missing data. The study data were presented along with the results of ITT analysis.

This study was approved by the Mersin University Ethical Committee of Clinical Research (approval number: 4/50, date: 23.02.2016) and by the Ethical Committee of Educational Unit of Mersin Public Hospitals Administration. All of the participants provided written informed voluntary consent. Participants were informed that their participation was voluntary, that they were free to quit the study without providing an excuse, that they could contact the researcher by phone as necessary, and that all of the collected data would be kept completely confidential and secured.

ELIGIBILITY:
Inclusion Criteria:

* expression of sleep problem,
* being literate,
* being able to communicate in Turkish,
* aged between 18-45 years old,
* being in the early postpartum period which lasts 2-6 weeks postpartum
* having delivered a single fetus with birth weight between 2500 and 4000 grams in the vertex presentation via a vaginal route,
* currently full breastfeeding

Exclusion Criteria:

* having experienced complications in the postpartum period (e.g., acute infections and fever states, history of myocardial infarction, irregular blood pressure, epilepsy, diabetes, osteoporosis, deep vein thrombosis, malignant melanoma, eclampsia, and/or preeclampsia),
* diabetic foot,
* open wound, varices, edema, or fungal infection in the foot,
* having been diagnosed with a psychiatric disorder (e.g., postpartum depression, psychosis, etc.), (
* undergoing pharmacological treatment for sleeplessness,
* alcohol intake

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-01; Primary Completion 2017-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Postpartum Sleep Quality Scale (PSQS) | The prettest data were collected on the 14th day.
  The items of the Postpartum Sleep Quality Scale are scored between 0 and 4 on a 5-point Likert scale (0 never, 4 always). Items 1, 2, and 14 are scored in reverse.To calculate the total score, subscale scores are collected. The minimum score of the The Postpartum Sleep Quality Scale is 0, and the maximum available score is 56. Higher PSQS scores indicate worse sleep quality .
sleep durations | The prettest data were collected on the 14th day.
  Personal Information Form

SECONDARY OUTCOMES:
Postpartum Sleep Quality Scale (PSQS) | The posttest data were collected on the 20th day.
  The items of the Postpartum Sleep Quality Scale are scored between 0 and 4 on a 5-point Likert scale (0 never, 4 always). Items 1, 2, and 14 are scored in reverse.To calculate the total score, subscale scores are collected. The minimum score of the The Postpartum Sleep Quality Scale is 0, and the maximum available score is 56. Higher PSQS scores indicate worse sleep quality .
sleep durations | The posttest data were collected on the 20th day.
  Personal Information Form

CONTACTS AND LOCATIONS:
Overall Officials: Nida SELVİ, Principal Investigator — Mersin University

IPD SHARING:
Plan to Share IPD: No